CLINICAL TRIAL: NCT01734746
Title: Sentinel Node Detection in Clinical Early Stage Ovarian Cancer
Acronym: SONAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL40323.068.12
Record Dates: First submitted 2012-10-31; First posted 2012-11-28 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-04

CONDITIONS: Ovarian Cancer; Sentinel Node
Keywords: ovarian cancer; sentinel node
MeSH Terms: conditions — Ovarian Neoplasms | interventions — technetium Tc 99m nanocolloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tracerinjection (Experimental): The intervention concerns tracerinjection (both blue dye and the radioactive isotope beingtechnetium-99-m-labeled albumin nanocolloid) in the ligamentum ovarii proprium (median side) and the ligamentum infundibulo-pelvicum (lateral side), close to the ovary and just below the peritoneum.
  Interventions: Procedure: Tracerinjection

INTERVENTIONS:
Procedure: Tracerinjection — The intervention concerns the tracerinjection for detection of the sentinel node.
  Other Names: 99mTc-nanocolloid or Nanocoll

SUMMARY:
As most cancers, ovarian cancer also spreads to regional lymph nodes. The concept of sentinel lymph node surgery is to see whether the cancer has spread to the very first lymph node or sentinel node (SN). If the sentinel node does not contain cancer, there is a high likelihood that the cancer has not spread to other lymph nodes. This means that, at least theoretically, a radical lymphadenectomy could be omitted and thus the associated morbidity. The sentinel node technique has been proven to be effective in different cancers such as breast cancer and malignant melanoma. In gynaecological tumors it has been shown to be effective in vulvar cancer. Currently sentinel node studies are done for cervix and uterine cancer.

The present study determines whether or not a sentinel node procedure in patients with ovarian cancer is feasible when the tracers are injected in the ovarian ligaments.

DETAILED DESCRIPTION:
According to the International Federation of Gynecology and Obstetrics (FIGO), Epithelial Ovarian Cancer (EOC) with lymph node metastases is classified as FIGO stage IIIC disease, even in the absence of peritoneal metastases. In contrast to patients with FIGO stage I ovarian cancer after a comprehensive staging procedure, patients with a FIGO stage III ovarian cancer obtain adjuvant chemotherapy. Therefore, the recognition of lymph node metastases is of utmost importance. In general, the incidence of lymph node metastases in clinical early stage EOC is approximately 14%, and depends on subtype histology (i.e. serous 23%, mucinous 3%) and differentiation grade (4% and 20% in grade 1 and 3 tumors respectively).

Surgical staging of EOC and the extent of lymph node dissection differs greatly from centre to centre. In case of a clinical early stage ovarian cancer, the Dutch guideline recommends a staging laparotomy with adequate lymph node sampling, with an absolute minimum of ten lymph nodes removed. In the same guideline, a footnote is made stating that a larger number of removed lymph nodes will increase the chance of finding metastases. These lymph nodes also need to be sampled from different anatomical regions, of which the most important are the para-aortic and paracaval region between the renal vein and inferior mesenteric artery, the common, internal and external iliac vessels and the obturator fossa.

A systematic lymphadenectomy can be seen as the golden standard. However, such a radical procedure gives more late morbidity than lymph node sampling. These include the formation of lymphocyst (up to 13.5%), nerve and vessel injury (up to 4%), and increased blood loss and operating time [26, 27]. Studies done for sentinel node in ovarian cancer are very limited and performed in women with uterine cancer by injecting the tracers in the ovary. In case of ovarian cancer such a procedure gives a possible risk of tumour dissemination. In this feasibility study the tracers are injected in the ligaments of the ovary, not in the cortex itself.

Patients with (suspicion of) ovarian cancer as well as patients with a high-grade uterine carcinoma will be included. The latter group of patients can also be included because these patients undergo the same surgical procedure; Total Abdominal Hysterectomy (TAH) with Bilateral Salpingo-Oophorectomy (BSO) and a pelvic and para-aortic lymphadenectomy or lymph node sampling.

Both blue dye and the radioactive isotope will be injected in the ligamentum ovarii proprium (median side) and the ligamentum infundibulo-pelvicum (lateral side), close to the ovary and just below the peritoneum.

In case of an ovarian tumor: after 15 minutes time-interval the ovarian mass will be removed and presented to the pathologist for a frozen section. If the result is benign, no further actions will be performed in these patients. If the result is malignant, the sentinel node(s) will be identified either by the radioactive tracer and / or visually (blue dye) after opening the retroperitoneal space. After removal of the sentinel node(s) a complete standard staging procedure will be performed including a comprehensive sampling of other lymph nodes at the different locations.

In case of endometrial cancer: after 15 minutes time-interval the surgical staging procedure starts with a TAH and BSO. After approximately 45 minutes the sentinel node(s) will be identified either by the radioactive tracer and / or visually (blue dye) after opening the retroperitoneal space. This 45 minutes time-interval is chosen to mimic the time interval when a frozen section is performed in case of an ovarian tumor. After removal of the sentinel node(s) a complete standard staging procedure will be performed including a comprehensive at random sampling of other lymph nodes at the different locations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a high suspicion of a malignant ovarian tumour planned for exploratory laparotomy.
* Patients with high-risk endometrial cancer in whom a staging laparotomy is planned.
* Age between 18 and 85 years.

Exclusion Criteria:

* Previous surgery of both ovaries.
* Previous vascular surgery of the aorta, caval vein, and/or iliac vessels.
* Previous lymphadenectomy of lymph node sampling in the iliac or para-aortal region.
* History of a malignant lymphoma.
* History of a malignant tumour in the abdominal cavity.
* Previous allergic reaction to blue dye.
* Pregnant or lactating patients.
* An allergy for human albumin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Kruitwagen, MD, PhD, Study Director — Maastricht UMC
Locations (1):
- MaastrichtUMC, Maastricht, Limburg, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Sentinel Node Procedure: Injection of both blue dye and the radioactive isotope (technetium-99-m-labeled albumin nanocolloid) in the ligamentum ovarii proprium (median side) and the ligamentum infundibulo-pelvicum (lateral side), close to the ovary and just below the peritoneum.
  blue dye and radioactive tracer
Period: Overall Study
Arm/Group | Sentinel Node Procedure
Started | 22
Completed | 21
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sentinel Node Procedure
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants] — Age (categorical) of participants at the time of surgery.;
  Participants
    <=18 years | 0
    Between 18 and 65 years | 12
    >=65 years | 10
Age, Continuous [Mean (Full Range); unit: years] — Ages (continuous) of participants at the time of surgery.
  years | 58.6 [22 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients (%) in Which Sentinel Node(s) Are Detected After Injection of Blue Dye and Tracer in the Ovarian Ligaments.
Time Frame: During surgery.
Population: see Kleppe et al., J Nucl Med 2014; 55:1799-1804
Measure: Number; unit: participants
Groups:
- Sentinel Node Procedure: Injection of both blue dye and the radioactive isotope (technetium-99-m-labeled albumin nanocolloid) in the ligamentum ovarii proprium (median side) and the ligamentum infundibulo-pelvicum (lateral side), close to the ovary and just below the peritoneum.
Arm/Group | Sentinel Node Procedure
Number analyzed (Participants) | 21
participants | 21

2. Secondary Outcome: Anatomical Location(s) of the Sentinel Nodes.
Description: The number of patients with only paraaortic/paracaval, only pelvic, and both paraaortic/paracaval and pelvic sentinel node locations.patients.
Time Frame: During surgery.
Measure: Number; unit: participants
Arm/Group | Sentinel Node Procedure
Number analyzed (Participants) | 21
participants
  SN only paraaortic | 14
  SN only pelvic | 2
  SN both paraortic and pelvic | 5

3. Other Pre Specified Outcome: Number of Patients With False Negative Sentinel Nodes.
Time Frame: During surgery.
Measure: Number; unit: participants
Arm/Group | Sentinel Node Procedure
Number analyzed (Participants) | 21
participants | 0

ADVERSE EVENTS:
Arm/Group | Sentinel Node Procedure
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2013-05-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT01734746/Prot_000.pdf